CLINICAL TRIAL: NCT00986414
Title: 13-week, Double-blind, Placebo-controlled, Fixed-dose, Multicenter Study to Evaluate the Efficacy and Safety of AFQ056 in Reducing Moderate to Severe L-dopa Induced Dyskinesias in Patients With Parkinson's Disease
Brief Title: Evaluation of the Efficacy and Safety of AFQ056 in Reducing Moderate to Severe L-dopa Induced Dyskinesias in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2208; EUDRACT number 2008-008712-98
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Parkinson Disease; Dyskinesias
Keywords: Parkinson Disease; L-dopa; Levodopa; dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- AFQ056-10mg (Experimental)
  Interventions: Drug: AFQ056
- AFQ056-25mg (Experimental)
  Interventions: Drug: AFQ056
- AFQ056-50mg (Experimental)
  Interventions: Drug: AFQ056
- AFQ056-75mg (Experimental)
  Interventions: Drug: AFQ056
- AFQ056-100mg (Experimental)
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056
  Arms: AFQ056-10mg
Drug: AFQ056
  Arms: AFQ056-25mg
Drug: AFQ056
  Arms: AFQ056-50mg
Drug: AFQ056
  Arms: AFQ056-75mg
Drug: AFQ056
  Arms: AFQ056-100mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This phase IIb study is designed to determine the safe and efficacious dose or dose range of AFQ056 for the treatment of patients with moderate to severe Parkinson's disease with L-Dopa induced dyskinesias.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with Parkinson's disease (PD), treated with L-Dopa, experiencing dyskinesias for at least three months

Exclusion Criteria:

* Surgical treatment for PD
* Cancer within the past 5 years (other than localized skin cancer and prostate cancer that has been effectively treated)
* Advanced, severe or unstable disease (other than PD) that may interfere with the study outcome evaluations

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in the modified AIMS (Abnormal Involuntary Movement Scale) total score | 12 weeks

SECONDARY OUTCOMES:
Disability due to dyskinesias as measured by change from baseline to endpoint in the PDYS-26 (26-Item Parkinson Disease Dyskinesia Scale) total score | 12 weeks
Change from baseline on patient's dyskinesia, disability caused by the dyskinesia and the underlying symptoms of PD as assessed by a clinician-rated (CGIC) and a patient-rated (PGIC) global impression of change | 12 weeks
Anti-dyskinetic efficacy as measured by items 32 and 33 of Part IV of the UPDRS (Unified Parkinson's Disease Rating Scale) | 12 weeks
Worsening of underlying symptoms of PD as measured by: UPDRS Part III; patient diary (dyskinesias); patient/clinician assessments of change in PD symptoms; AEs related to worsening of PD | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- Australia (5):
  - Novartis Investigative Site, East Gosford
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Melbourne
  - Novartis Investigative Site, Parkville
  - Novartis Investigational Site, Westmead
- Canada (7):
  - Quebec Memory & Motor Skills Disorders Clinic, Québec, Quebec
  - Clinique Neuro-Outaouais, Gatineau
  - Recherches Pembina, Inc, Greenfield Park
  - Novartis Investigative Site, Montreal
  - Parkinson's and Neurodegenerative Disorders Clinic, Ottawa
  - Toronto Western Hospital, UHN, Toronto
  - Novartis Investigative Site, Vancouver
- Finland (5):
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Lahti
  - Novartis Investigative Site, Oulu
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (5):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulouse
- Germany (9):
  - Novartis Investigative Site, Beelitz-Heilstätten
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Tübingen
- Italy (3):
  - Novartis Investigative Site, Lido di Camaiore
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Roma
- Japan (6):
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative SIte, Tokyo
  - Novartis Investigative Site, Tōon
  - Novartis Investigative Site, Wakayama
- Spain (3):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Madrid

REFERENCES:
- [Result] Stocchi F, Rascol O, Destee A, Hattori N, Hauser RA, Lang AE, Poewe W, Stacy M, Tolosa E, Gao H, Nagel J, Merschhemke M, Graf A, Kenney C, Trenkwalder C. AFQ056 in Parkinson patients with levodopa-induced dyskinesia: 13-week, randomized, dose-finding study. Mov Disord. 2013 Nov;28(13):1838-46. doi: 10.1002/mds.25561. Epub 2013 Jul 12. PMID 23853029